CLINICAL TRIAL: NCT03333993
Title: Randomized Trial With Mat Pilates in Women With Breast Cancer During Adjuvant Radiotherapy
Brief Title: Mat Pilates in Women With Breast Cancer During Adjuvant Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 64099717.7.0000.5274
Record Dates: First submitted 2017-10-31; First posted 2017-11-07 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Adjuvant Radiotherapy
Keywords: Pilates exercise; Fatigue; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in this group will be submitted to 10 sessions of Mat Pilates exercises, performed twice a week, lasting 60 minutes, for a period of 5 weeks (from the beginning to the end of radiotherapy). The program will consist of group sessions of up to 4 patients, supervised by a specialized physiotherapist. In addition, they will be guided to follow with the home exercises, according to the institutional routine.
  Interventions: Other: Pilates Exercise; Other: Home exercises
- Control Group (Active Comparator): Patients assigned to this group will not participate in the Mat Pilates exercises and will be instructed to maintain the home exercises for upper limbs, guided by physiotherapists in the postoperative period, according to the institutional routine.
  Interventions: Other: Home exercises

INTERVENTIONS:
Other: Pilates Exercise — The Mat Pilates exercise will be performed twice a week and the duration of the sessions will be 60 minutes, consisting of 5 minutes of warm-up exercises, 50 minutes of strengthening exercises followed by 5 minutes of relaxation and stretching.
  Other Names: Pilates method
  Arms: Intervention Group
Other: Home exercises — Exercises for upper limbs according to the institutional routine.
  Other Names: Institutional Routine

SUMMARY:
Breast cancer is the most frequent tumor site among women in the world (FERLAY et al., 2015). In Brazil, estimates for the year 2017 indicate the occurrence of about 57,960 new cases (56.2 cases per 100,000 women); (Brazil - Ministry of Health, 2015). The increase in adjuvant therapies resulted in an estimated increase of 22 million cancer survivors worldwide (GOLDSTEIN et al., 2012). However, as survival rates increased, more women faced complications related to diagnosis and treatment (ABRAHMS et al., 2016). Adjuvant radiotherapy is a frequent treatment in breast cancer and fatigue it is the main adverse effects (HICKOK et al., 2005). Measures of intervention through physical activity have shown benefits in the increase of the functional capacity that generates a reduction of effort and decrease of the fatigue (MARKES et al., 2009). General Objective: To evaluate the influence of Mat Pilates on fatigue, quality of life, functional capacity, flexibility, lymphedema, radiodermatitis and depression, in the women with breast cancer and with an indication of adjuvant radiotherapy, at the Cancer Hospital III of the National Cancer Institute (INCA). After recruitment, women will be allocated randomly in: Intervention Group (Mat Pilates and usual activities) and Control Group (usual activities). Patients in the intervention group will be submitted to 10 sessions of Mat Pilates for a period of 5 weeks (from beginning to end of adjuvant radiotherapy). Patients assigned to the control group will not participate in the Mat Pilates program, but will maintain the usual exercises for upper limbs, guided by physiotherapists in the postoperative period. In both groups, patients will be submitted, functional capacity assessment, flexibility assessment, assessment of the presence of lymphedema, and questionnaire application of fatigue, quality of life, level of physical activity and depression. Will be performed a descriptive analysis of the population. Univariate logistic regression will be performed between the outcomes according to the exercise groups and also, for the possible confounding variables. The variables with p<0.20 will be selected for adjustment in the construction of the multiple logistic regression model. Those with p<0.05 and/or with clinical significance will be maintained in the model.

DETAILED DESCRIPTION:
After recruitment, women will be randomly assigned to: Intervention Group (Mat Pilates and usual activities) and Control Group (usual activities). At patients in the intervention group will be submitted to 10 sessions of Mat Pilates for a period of 5 weeks (from beginning to end of adjuvant radiotherapy). The Mat Pilates program will be based on group sessions with the supervision of physiotherapists specialized in technique. The groups will consist of a maximum of 4 patients, to achieve the basic principles of the technique that include concentration, control, accuracy and fluidity of movement. Mat Pilates sessions will be held in the physiotherapy gymnasium of Cancer Hospital III / INCA. The Mat Pilates program will be held twice a week and the duration of sessions will be 60 minutes, consisting of 5 minutes of exercises 50 minutes of strengthening exercises with flexibilization of the muscular fibers, where the concentric phase of the movement will be performed at the expiration, followed by 5 minutes of relaxation and stretching. The movements will be carried out slowly and with the maximum of 2 sets of 10 replicates. The Swiss ball and elastic band accessories will be used. The Mat Pilates intensity exercises will be controlled by means of the adapted Borg Scale (0-10), where the perception of the effort will vary from 2 (very light) to 7 (moderate-intense). On days of the week in which the patient will not practice the Mat Pilates program, the usual upper limb exercises will be maintained by the physiotherapists on the first postoperative day at Cancer Hospital III / INCA. Patients allocated to the control group will not participate in the Mat Pilates program, but will be directed to maintain the usual exercises for upper limbs, guided by physiotherapists in the postoperative. In both groups, the patients will be submitted, the functional capacity evaluation composed of the Disability Arm, Shoulder and Hand (DASH) questionnaire, flexibility assessment, presence of lymphedema, radiodermatitis and application of the questionnaires International Questionnaire of Physical Activity (IPAQ), Functional Assessment of Cancer Therapy- Fatigue (FACT-F) for Fatigue, European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core-30 (EORTC QLQ-C30) and specific module EORTC QLQ Breast-23 (EORTC QLQ-BR23) for quality of life, and Geriatric Depression Scale(GDS) for depression at the time of study inclusion and in the follow-up (end of radiotherapy, 30 days and 6 months after end).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older
* Women with indication of adjuvant radiotherapy in the period from March 15, 2017 to May 30, 2019 to be performed exclusively at the Hospital de Cancer III (INCA / HCIII).

Exclusion Criteria:

* Women who practice physical activity at least 2 times a week for 1 hour
* Women with previous cancer diagnosis
* Women submitted to immediate breast reconstruction
* Presence of acute infections and orthopedic, neurological, decompensated cardiorespiratory and severe renal dysfunction
* Women who are not able to respond to questionnaires and not to agree to sign the Informed Consent Form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Fatigue | 2 years
  It will be assessed by FACIT-FATIGUE (Version 4) questionnaire.

SECONDARY OUTCOMES:
Quality of Life in breast cancer | 2 years
  It will be measured by EORTC QLQ - BR23 questionnaire.
Functionality | 2 years
  It will be evaluated by Brazilian DASH questionnaire.
Depression | 2 years
  This outcome will be measured by GDS-15 questionnaire.
Quality of life related to health | 2 years
  It will be measured by EORTC QLQ- C30 questionnaire.
Physical activity level | 2 years
  It will be measured by IPAQ questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Torres, master, Principal Investigator — National Cancer Institute, France
Locations (1):
- Daniele Medeiros Torres, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Torres DM, de Menezes Fireman K, Fabro EAN, Thuler LCS, Koifman RJ, Bergmann A, da Silva Santos S. Effectiveness of mat pilates on fatigue in women with breast cancer submitted to adjuvant radiotherapy: randomized controlled clinical trial. Support Care Cancer. 2023 May 30;31(6):362. doi: 10.1007/s00520-023-07824-1. PMID 37249715